CLINICAL TRIAL: NCT01680861
Title: Randomized, Open-Label Trial of Tacrolimus/Everolimus vs. Tacrolimus/Enteric-Coated Mycophenolate Sodium to Prevent Biopsy-Proven Acute Rejection and Chronic Allograft Injury in Adult, Primary Kidney Transplantation
Brief Title: Tacrolimus/Everolimus Versus Tacrolimus/Enteric-Coated Mycophenolate Sodium
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gaetano Ciancio (Other)
Responsible Party: Sponsor-Investigator, Gaetano Ciancio, Professor of Surgery, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20110126
Record Dates: First submitted 2012-03-06; First posted 2012-09-07 (Estimated); Results first posted 2016-12-15 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-10

CONDITIONS: Transplant; Failure, Kidney
Keywords: Kidney transplant patients
MeSH Terms: interventions — Tacrolimus; Everolimus; Mycophenolic Acid; Adrenal Cortex Hormones; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus and Everolimus (Experimental): Patients in both arms will receive reduced tacrolimus dosing (rTd), 0.1 mg/kg PO divided in two daily doses - beginning when serum Cr decreases to a level of <4 mg/dl (i.e., acceptable renal transplant function) postoperatively. Target tacrolimus trough levels during the first year post-transplant and thereafter will be 5-8 ng/ml.
  Everolimus initiated within 24 hours post-transplant (i.e., immediately following randomization) at 0.75mg PO BID and will be adjusted in order to achieve target everolimus trough levels of 3-8 ng/ml.
  Interventions: Drug: Tacrolimus; Drug: Everolimus; Drug: Corticosteroids
- Tacrolimus and Enteric-Coated Mycophenolate Sodium (EC-MPS) (Active Comparator): Patients in both arms will receive reduced tacrolimus dosing (rTd), 0.1 mg/kg PO divided in two daily doses - beginning when serum Cr decreases to a level of <4 mg/dl (i.e., acceptable renal transplant function) postoperatively. Target tacrolimus trough levels during the first year post-transplant and thereafter will be 5-8 ng/ml.
  EC-MPS will be initiated at 720 mg PO BID starting on the first post-operative day.
  Interventions: Drug: Tacrolimus; Drug: Enteric Coated Mycophenolate Sodium (EC-MPS); Drug: Corticosteroids

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus dosing (rTd) is planned, 0.1 mg/kg PO BID - beginning when serum Cr decreases to a level of <4 mg/dl (i.e., acceptable renal transplant function) postoperatively. Target tacrolimus trough levels during the first year post-transplant and thereafter will be 5-8 ng/ml.
  Other Names: Prograf (brand name)
Drug: Everolimus — Everolimus initiated at 0.75 PO BID and will be adjusted in order to achieve target everolimus trough levels of 3-8 ng/ml.
  Other Names: Zortress (brand name)
  Arms: Tacrolimus and Everolimus
Drug: Enteric Coated Mycophenolate Sodium (EC-MPS) — EC-MPS 720 mg PO BID - beginning on 1st postoperative day.
  Other Names: Myfortic (brand name)
  Arms: Tacrolimus and Enteric-Coated Mycophenolate Sodium (EC-MPS)
Drug: Corticosteroids — Corticosteroids will be given as per our center protocol, i.e., a bolus of 500 mg of Methylprednisolone intravenously at surgery and daily x2, followed by 1.0 mg/kg, then 0.5 mg/kg orally until weaned off completely by 7-10 days postoperatively - the plan is for corticosteroids to be discontinued by 7-10 days postoperatively in both groups.
  Other Names: Methylprednisolone

SUMMARY:
A recent therapeutic strategy following renal transplantation includes simultaneous use of reduced calcineurin inhibitor (CNI) dosing and maximized use of a non-nephrotoxic, antiproliferative drug (inosine monophosphate dehydrogenase (IMPDH) or TOR inhibitor), with the goals of reducing/avoiding CNI nephrotoxicity, the incidence of acute rejection, and chronic allograft injury (CAI) (i.e., interstitial fibrosis/tubular atrophy), leading to more favorable longer-term patient and graft survival.1-7 Early corticosteroid withdrawal has also been used in the attempt to avoid well-known side effects while maintaining favorable patient and graft survival.8-10 While the investigators center and numerous other centers have also included single agent, antibody induction utilizing the lymphodepleting polyclonal antibody rabbit anti-human thymocyte globulin (ATG), nondepleting human anti-interleukin-2 receptor (CD25) monoclonal antibody daclizumab (Dac) or basiliximab, or lymphodepleting humanized anti-CD52 monoclonal antibody alemtuzumab,11-17 evidence now suggests that an even more effective induction strategy may include the combined use of more than one induction agent (each with fewer doses than if used alone), with the goal of bringing the kidney transplant recipient even closer (through more effectively timed lymphodepletion) to an optimally immunosuppressed state, allowing further reduction in long-term maintenance drug dosing.18-25 The investigators have now successfully used dual ATG/Dac induction therapy in both kidney-alone23-24 and simultaneous kidney-pancreas (SPK) transplantation,18-20 and a recent report from the investigators center of kidney-alone and SPK recipients shows that the addition of anti-CD25 to ATG for induction therapy more effectively delays the return of peripheral blood CD25+ cells.25 In the kidney-alone recipient study 3 doses of ATG were combined with 2 doses of Dac for induction,23-24 vs. the investigators previous studies utilizing single agent induction with 7 doses of ATG or 5 doses of Dac.4,16,17 Successful combination of ATG/basiliximab as dual induction in kidney transplantation has also been reported elsewhere,21-22 along with equivalency in clinical outcomes using daclizumab vs. basiliximab.13

DETAILED DESCRIPTION:
A. Primary Objectives:

1. The percentage of patients who develop chronic allograft injury (CAI) progression during the first 12 months post-transplant protocol biopsy (i.e., higher grade of IF/TA at either the 6 or 12 month protocol biopsy in comparison with the baseline biopsy).
2. The incidence rate of biopsy-proven acute rejection (BPAR) during the first 12 months post-transplant.

B. Secondary Objectives:

1. Adverse events including graft loss (death-censored and death-uncensored), and death at 12 months post-transplant.
2. Incidence rate and severity (severity of CAI at 12 months as well), based upon careful review of all clinically indicated and protocol biopsies.
3. Renal function as determined by serum creatinine and estimated glomerular filtration rate (eGFR) (calculated using the abbreviated MDRD formula) at 12, months post-transplant. Use of multivariable analysis to compare renal function as well as BPAR and CAI progression will also be performed (particularly, after adjusting for the significant effects of donor age, recipient age, race/ethnicity, and any other predictors).

5. Adverse events including withholding (for ≥ 28 days) or discontinuance of study medications (and reasons why), new onset diabetes mellitus after transplantation (NODAT), infections requiring hospitalization, and requirement of anti-lipid medication at 12 months post-transplant.

6. Avoidance of the requirement for maintenance corticosteroid therapy after renal transplantation.

7. Allowance of reduced maintenance tacrolimus dosing (rTd).

ELIGIBILITY:
Inclusion Criteria:

* Weight > 40 kg.
* Deceased donor (SCD) or LD.
* Donor-recipient 1 haplotype matched pairs with a minimum matching of 1 HLA DR antigen.
* Negative standard cross match for T cells.
* Pretransplant panel reactive antibodies of < 30%.
* Graft required to be functional, producing at least 100ml of urine within 24hr after transplantation.

Exclusion Criteria:

* Previously received or is receiving an organ transplant other than a kidney.
* Donor organ with a cold ischemic time > 48 hours.
* ABO incompatible donor kidney.
* Recipients of T cell, or B cell crossmatch positive transplant.
* Panel reactive antibody (PRA) >30%
* HIV or Hepatitis C virus, or Hepatitis B virus antigenemia.
* Current malignancy or a history of malignancy
* Liver disease
* Uncontrolled concomitant infections and/or severe diarrhea, vomiting, active upper gastro-intestinal tract malabsorption or an active peptic ulcer
* Use of warfarin, fluvastatin, or herbal supplements during the study.
* Use of astemizole, pimozide, cisapride, terfenadine, or ketoconazole.
* Hypersensitivity to thymoglobulin, IL-2 receptor inhibitor monoclonal antibodies, tacrolimus, everolimus, MPA, or corticosteroids.
* Pregnant or lactating.
* Abnormal screening/baseline labs WBC, platelet count, triglycerides, and cholesterol Double kidneys,ECD, pediatric en-block, and donation after cardiac death (DCD)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Ciancio, M.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Tacrolimus/Everolimus: our experimental maintenance arm: Target 12-hr Tacrolimus trough level: 5-8 ng/mL Target 12-hr Everolimus trough level: 3-8 ng/mL.
- Tacrolimus/EC-MPS: our standard maintenance arm: Target 12-hr Tacrolimus trough level: 5-8 ng/mL Target EC-MPS dose: 720 mg PO BID (as tolerated).
Period: Early Post-transplant Period
Arm/Group | Tacrolimus/Everolimus | Tacrolimus/EC-MPS
Started | 16 (One patient didn't produce sufficient urine during first 24hr post-transplant (ineligible).) | 16 (One patient developed immediate DGF (delayed graft function) and was therefore ineligible.)
Completed | 15 | 15
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1
Period: First 12 Months Post-transplant
Arm/Group | Tacrolimus/Everolimus | Tacrolimus/EC-MPS
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tacrolimus/Everolimus: our experimental maintenance arm.
- Tacrolimus/EC-MPS: our standard maintenance arm.
- Total: Total of all reporting groups
Arm/Group | Tacrolimus/Everolimus | Tacrolimus/EC-MPS | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (10.5) | 48.5 (11.2) | 49.2 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 12 | 11 | 23
Race/Ethnicity, Customized [Number; unit: participants]
  African-American | 5 | 2 | 7
  Hispanic | 7 | 10 | 17
  White/Asian | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: BPAR (Biopsy-proven Acute Rejection) Incidence During the First 12 Months Post-transplant
Description: BPAR (biopsy-proven acute rejection) incidence during the first 12 months post-transplant. Grading is determined using standard Banff criteria.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Tacrolimus/Everolimus | Tacrolimus/EC-MPS
Number analyzed (Participants) | 15 | 15
participants | 1 | 3
Statistical Analysis 1: Comparison: Tacrolimus/Everolimus vs Tacrolimus/EC-MPS; Test type: Superiority or Other; p = 0.32, Log Rank

2. Secondary Outcome: Incidence of Chronic Allograft Nephropathy (CAI) at 12 Months Post-transplant
Description: Incidence of (biopsy-proven) chronic allograft nephropathy (CAI) [interstitial fibrosis and tubular atrophy, using standard Banff criteria] at 12 months post-transplant.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Tacrolimus/Everolimus | Tacrolimus/EC-MPS
Number analyzed (Participants) | 15 | 15
participants | 3 | 3
Statistical Analysis 1: Comparison: Tacrolimus/Everolimus vs Tacrolimus/EC-MPS; Test type: Superiority or Other; p = 0.99, Log Rank

3. Secondary Outcome: Graft Loss (Return to Permanent Dialysis or Death)
Time Frame: during the first 12 months post-transplant
Measure: Number; unit: participants
Arm/Group | Tacrolimus/Everolimus | Tacrolimus/EC-MPS
Number analyzed (Participants) | 15 | 15
participants | 0 | 0
Statistical Analysis 1: Comparison: Tacrolimus/Everolimus vs Tacrolimus/EC-MPS; Test type: Superiority or Other; p = 1.0, Log Rank

4. Secondary Outcome: eGFR (Calculated Glomerular Filtration Rate), i.e., Renal Function, at 1 Month Post-transplant.
Description: using the abbreviated MDRD formula.
Time Frame: at 1 month post-transplant
Measure: Mean (Standard Error); unit: ml/min per 1.73 m2
Arm/Group | Tacrolimus/Everolimus | Tacrolimus/EC-MPS
Number analyzed (Participants) | 15 | 15
ml/min per 1.73 m2 | 82.1 (8.2) | 62.1 (6.2)
Statistical Analysis 1: Comparison: Tacrolimus/Everolimus vs Tacrolimus/EC-MPS; Test type: Superiority or Other; p = 0.06, t-test, 2 sided

5. Secondary Outcome: eGFR (Renal Function) at Month 3 Post-transplant
Description: Renal function as determined by the estimated glomerular filtration rate (eGFR) at 3 months post-transplant, using the abbreviated MDRD formula.
Time Frame: at 3 months post-transplant
Measure: Mean (Standard Error); unit: ml/min per 1.73 m^2
Arm/Group | Tacrolimus/Everolimus | Tacrolimus/EC-MPS
Number analyzed (Participants) | 15 | 15
ml/min per 1.73 m^2 | 75.7 (6.0) | 65.6 (4.2)
Statistical Analysis 1: Comparison: Tacrolimus/Everolimus vs Tacrolimus/EC-MPS; Test type: Superiority or Other; p = 0.18, t-test, 2 sided

6. Secondary Outcome: eGFR (Renal Function) at 6 Months Post-transplant
Description: using the abbreviated MDRD formula.
Time Frame: at 6 months post-transplant
Measure: Mean (Standard Error); unit: ml/min per 1.73 m2
Arm/Group | Tacrolimus/Everolimus | Tacrolimus/EC-MPS
Number analyzed (Participants) | 13 | 14
ml/min per 1.73 m2 | 66.7 (5.0) | 63.7 (3.9)
Statistical Analysis 1: Comparison: Tacrolimus/Everolimus vs Tacrolimus/EC-MPS; Test type: Superiority or Other; p = 0.65, t-test, 2 sided

7. Secondary Outcome: Discontinuance of Any Study Medication (Tacrolimus, Everolimus, or EC-MPS)
Time Frame: during the first 12 months post-transplant
Population: Note: one patient in the Tacrolimus/EC-MPS arm discontinued EC-MPS at 12 months post-transplant following a colon cancer diagnosis and the necessity to receive chemotherapy.
Measure: Number; unit: participants
Arm/Group | Tacrolimus/Everolimus | Tacrolimus/EC-MPS
Number analyzed (Participants) | 15 | 15
participants | 0 | 1

ADVERSE EVENTS:
Time Frame: during the first 12 months post-transplant,
Description: Here, we are reporting the numbers of patients who 1) developed an infection requiring hospitalization (or had an opportunistic viral infection not requiring hospitalization) and 2) developed NODAT (new onset diabetes after transplant) (among patients not having pretransplant diabetes mellitus) during the first 12 months post-transplant. Please note that adverse events specified to be studied as secondary outcomes were the only AEs collected in our randomized trial.
Arm/Group | Tacrolimus/Everolimus | Tacrolimus/EC-MPS
Serious Adverse Events (participants affected / at risk) | 4/15 | 4/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus/Everolimus (N=15) | Tacrolimus/EC-MPS (N=15)
Urinary Tract Infection Requiring Hospitalization (Infections and infestations) | 1 (1) | 0 (0)
Ear Infection Requiring Hospitalization (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
CMV Viremia (Infections and infestations) | 0 (0) | 1 (1)
Polyoma Viral Infection (Viremia) (Infections and infestations) | 2 (2) | 1 (1)
Herpes Zoster Infection (Infections and infestations) | 1 (1) | 0 (0)
NODAT (Endocrine disorders) | 2 (2) | 0 (0) — Occurrence of New Onset Diabetes after Transplant among patients not having pretransplant diabetes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No